CLINICAL TRIAL: NCT00947752
Title: An Open-Label, Multicenter, Randomized Study Evaluating the Tolerability and Safety of Two Formulations of Glatiramer Acetate (GA) for Subcutaneous Injection
Brief Title: Safety of New Formulation of Glatiramer Acetate
Acronym: Song
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PM033
Record Dates: First submitted 2009-07-25; First posted 2009-07-28 (Estimated); Results first posted 2011-06-09 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis (RRMS); Glatiramer Acetate (GA)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- F1 Glatiramer acetate 20mg/1.0ml (Active Comparator)
  Interventions: Drug: Glatiramer Acetate
- F2 Glatiramer acetate 20mg/0.5ml (Experimental)
  Interventions: Drug: Experimental Glatiramer Acetate

INTERVENTIONS:
Drug: Glatiramer Acetate — Subjects received both doses once daily in a crossover fashion, for a total treatment duration of five weeks, including a one-week run-in period. Subject-reported injection pain was recorded in a daily diary.
  Other Names: F1
  Arms: F1 Glatiramer acetate 20mg/1.0ml
Drug: Experimental Glatiramer Acetate — GA 20 mg/0.5 mL
  Other Names: F2
  Arms: F2 Glatiramer acetate 20mg/0.5ml

SUMMARY:
The purpose of this study is to compare pain associated with injections and injection-site reactions of the approved formulation of Glatiramer Acetate (GA) versus investigational formulation of GA. In addition, the investigators will evaluate the side effects of the two formulations of GA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age with a diagnosis of RRMS
* Currently injecting GA 20mg/1.0mL per day subcutaneously (SC) for a minimum of 90 days utilizing the autoject®2 for glass syringe or by a manual injection technique
* Willing to switch from autoject®2 for glass syringe to manual injection technique or continue with a manual injection technique during the course of the study
* Willing and able to be trained on a seven site injection rotation. Subject must be willing to comply with a minimum five injection site rotation plan during the study
* Willing and able to complete all procedures and evaluations related to the study
* Willing to continue to follow usual injection site preparation and routine adjunctive LISR management techniques
* Willing and able to provide written informed consent

Exclusion Criteria:

* Currently using or treated with another immunomodulating therapy (IMT) in conjunction with GA in the 30 days prior to screening for this study
* Currently using intermittent or pulse courses of corticosteroids by any route of administration in the 30 days prior to screening for this study. (Corticosteroids are prohibited for the duration of the study.)
* Currently using an investigational drug or using treatment with any other investigational agent in the 30 days prior to screening for this study
* Presence or history of skin necrosis
* Known extensive dermatological condition that could be a confounding factor
* Pregnant or planning pregnancy or breastfeeding
* Any physical condition that impairs ability to be injected at the minimum of five sites rotation
* Not able or willing to complete a daily diary
* Use of any other parenteral medications (e.g., intramuscular, SC, intravenous, etc.) either currently or in the past 30 days prior to screening for this study
* Any other medical or psychiatric conditions that would make the subject unsuitable for this research, as determined by the Investigator
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Smith, MD, Study Director — Teva Neuroscience, Inc.

REFERENCES:
- See also: Visual Analog Scale definition — http://en.wikipedia.org/wiki/Visual_analogue_scale

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomly assigned in a 1:1 assignment ratio to one of two drug sequences. Subjects were to manually inject GA (F1 or F2) once daily for 14 days then cross-over to the other formulation for another 14 days of treatment, including a 7-day run-in period on F1 treatment for all participants to assess daily diary compliance.
Pre-assignment Details: To ensure the standardization, all study sites were instructed to train subjects to complete the daily diary, with special attention to the Visual Analog Scale (VAS) used to measure pain.
Period: 7-Day Run-in Treatment Period
Arm/Group | F1 Glatiramer Acetate 20mg/1.0ml | F2 Glatiramer Acetate 20mg/0.5ml
Started | 147 (All subjects started with a daily does of F1 for 7 days) | 0
Completed | 147 | 0
Not Completed | 0 | 0
Period: 1st 14-day Treatment Period
Arm/Group | F1 Glatiramer Acetate 20mg/1.0ml | F2 Glatiramer Acetate 20mg/0.5ml
Started | 76 | 71
Completed | 76 | 71
Not Completed | 0 | 0
Period: Crossover to 2nd 14-day Treatment Period
Arm/Group | F1 Glatiramer Acetate 20mg/1.0ml | F2 Glatiramer Acetate 20mg/0.5ml
Started | 71 | 76
Completed | 71 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | F1 Glatiramer Acetate (GA) 20mg/1.0ml | F2 Glatiramer Acetate 20mg/0.5ml | Total
Number analyzed (Participants) | 76 | 71 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 71 | 144
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (10.64) | 46.9 (9.64) | 46.0 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 58 | 119
  Male | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Subject-reported Pain Associated Immediately After Each Injection
Description: A visual analog scale (VAS) was used for subjective characteristics that cannot be directly measured. Respondents specified their level of agreement to a statement by indicating a position along a continuous line between two end-points. The VAS scale used 0 mm to represent "no pain" and up to 100 mm to represent "worst possible pain;" subjects drew a continuous line to represent their level of pain.
Time Frame: 5 weeks of injections
Population: Of the 147 subjects to be analyzed, 3 were excluded for discontinuations due to withdraw of consent.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | F1 Glatiramer Acetate (GA) 20mg/1.0ml | F2 Glatiramer Acetate 20mg/0.5ml
Number analyzed (Participants) | 144 | 144
Scores on a scale | 11.89 (14.325) | 8.64 (10.825)

2. Secondary Outcome: Degree of Pain Within 5 Mins After Injection
Description: as for outcome 1
Time Frame: 5 weeks of injections
Population: Of the 147 subjects to be analyzed, 3 were excluded for discontinuations due to withdraw of consent.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | F1 Glatiramer Acetate (GA) 20mg/1.0ml | F2 Glatiramer Acetate 20mg/0.5ml
Number analyzed (Participants) | 144 | 144
Scores on a scale | 17.19 (18.583) | 11.85 (14.112)

ADVERSE EVENTS:
Arm/Group | F1 Glatiramer Acetate (GA) 20mg/1.0ml | F2 Glatiramer Acetate 20mg/0.5ml
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/147
Other Adverse Events (participants affected / at risk) | 0/147 | 0/147

LIMITATIONS AND CAVEATS:
Blinding in this study was not possible due to the subjects' ability to detect difference in the volume of each formulation. The lack of blinding was a known limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.